CLINICAL TRIAL: NCT06590415
Title: Trancriptomics and Lipidomics of Epicardial Ectopic Fat
Acronym: GENTLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM24_0060
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T2D/DGE patients (Experimental): Diagnostic age of diabètes mellitus less than or equal to 40 years and epicardial fat volume greater than 72 mL.
  Interventions: Procedure: Subcutaneous adipose tissue biopsy; Other: Blood sampling
- Control patients (Active Comparator): Age at diagnosis of diabetes greater than 40 and/or epicardial fat volume less than 72 mL.
  Interventions: Procedure: Subcutaneous adipose tissue biopsy; Other: Blood sampling

INTERVENTIONS:
Procedure: Subcutaneous adipose tissue biopsy — Under local anesthesia, subcutaneous adipose tissue will be collected from 2 puncture points in the umbilical region for a total volume of 2 mL.
Other: Blood sampling — One 4 mL tube of blood will be collected

SUMMARY:
Cohort studies have shown that patients with obesity associated with metabolic abnormalities (metabolically unhealthy obesity) have an accumulation of ectopic fat deposits (EDF) linked to subcutaneous adipose tissue dysfunction. Although it is accepted that the storage capacity of subcutaneous adipose tissue is genetically determined, the genetic factors predisposing to adipose tissue distribution abnormalities remain poorly understood.

The Angiosafe T2D cohort consists of 7200 highly phenotyped type 2 diabetes (T2D) patients. In 297 patients from this cohort (ancillary study), investigators assessed epicardial fat volume (EFV) using an artificial intelligence algorithm. In 42 of these patients, designated as early T2DM/DGE, an accumulation of epicardial fat and diabetes occurring before the age of 40 were observed, clinically approaching the clinical presentation of genetic lipodystrophy, although subcutaneous adipose tissue persisted in their case.

This study will focus on a case-control study nested within the pre-existing cohort of T2D patients (Angiosafe T2D), and more specifically within this cohort on a subgroup of 42 patients with early-onset diabetes and an abnormal distribution of adipose tissue caracterized by ectopic fat accumulation. In order to understand the severe metabolic phenotype observed in this group of 42 patients, investigators propose to perform a multiomic analysis combining clinico-biological, exomic, transcriptomic and lipidomic data.

This study will compare the rate of patients with at least one rare (<1% general population) potentially pathogenic genetic variant in a coding region of the genetic lipodystrophy genes by whole exome sequencing in 42 early-onset T2DM and a high epicardial fat volume patients versus 42 patients without early-onset T2DM and/or high epicardial fat volume (control group).

ELIGIBILITY:
Inclusion Criteria for T2D/DGE patient:

* Adult patient of legal age included in the Angiosafe T2D multicenter study, having consented to the use of the data collected for research purposes.
* Patient who has signed the GENTLE informed consent form.
* Patient not objecting to re-use of data and samples collected in the Angiosafe T2D study
* Patient with type 2 diabetes according to ADA recommendations
* Age at diagnosis of diabetes less than or equal to 40 years and epicardial fat volume greater than 72 mL*.
* Patient beneficiary or affiliated to a social security scheme

Inclusion Criteria for control patient:

* Adult patient of legal age included in the Angiosafe T2D multicenter study, having consented to the use of the data collected for research purposes.
* Patient who has signed the GENTLE informed consent form.
* Patient not objecting to re-use of data and samples collected in the Angiosafe T2D study
* Patient with type 2 diabetes according to ADA recommendations
* Age at diagnosis of diabetes greater than 40 and/or epicardial fat volume less than 72 mL
* Patient beneficiary or affiliated to a social security scheme

Exclusion Criteria:

* Type 1 diabetic patient
* Patient with monogenic diabetes
* Patient with diabetes secondary to pancreatic disease
* Pregnant or breast-feeding women, patients under guardianship, deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of variants genes | Day 1
  Higher frequency of rare heterozygous missense variants of lipodystrophy genes, or the presence of variants more often classified as pathogenic or of unknown significance (according to the ACMG classification) in the target group compared with the control group.
  A variant is considered rare if its frequency in GnomAD is < 1%.

SECONDARY OUTCOMES:
Plasma and adipocyte lipidic profil determined by mass spectrometry | Day 1
  Identification of plasma and adipocyte lipid species whose expression is significantly altered in patients according to their phenotype and genotype (T2D/DGE versus controls)
Integrative multiomic analysis including clinical, biological, exomic, transcriptomic and lipidomic data. | Day 1
  identification of a multiomic signature that would differentiate the 2 groups: Early T2D/DGE and controls.
Gene expression profil in subcutaneous adipose tissue determined by mRNA sequencing | Day 1
  identification of genes whose expression is significantly altered in patients according to their phenotype and genotype (comparison of early T2D/DGE versus controls) in subcutaneous adipose tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France